CLINICAL TRIAL: NCT03731234
Title: Phase II Multicenter Single Arm Study to Evaluate the Efficacy and Safety of Ibrutinib in Combination to Rituximab-CHOP Followed by Ibrutinib Maintenance in Untreated Patients With Activated-B-Cell (ABC)-DLBCL at Intermediate-high and High Risk (IPI ≥2)
Brief Title: Ibrutinib + R-CHOP Followed by Ibrutinib Maintenance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_RI-CHOP
Record Dates: First submitted 2018-10-04; First posted 2018-11-06 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: DLBCL
Keywords: DLBCL; Activated-B-Cell DLBCL; Ibrutinib; Phase II
MeSH Terms: interventions — ibrutinib

STUDY DESIGN:
Intervention Model Description: Ibrutinib in combination to rituximab-CHOP followed by ibrutinib maintenance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibrutinib+R-CHOP (Experimental): Screening phase for selection of Activated-B-Cell (ABC)-DLBCL Induction phase: R-CHOP21 x 5 cycles in combination with ibrutinib Maintenance phase: maintenance with Ibrutinib for 18 months for patients responding to the induction phase (CR or PR)
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib in combination to rituximab-CHOP followed by ibrutinib maintenance
  Other Names: IMBRUVICA (commercial name)

SUMMARY:
This is a prospective, multicenter, single arm, phase II trial in patients with ≥ 18 and <65 years with poor-prognosis (IPI ≥ 2) and newly diagnosed ABC-DLBCL.

Aim of the study is to assess the efficacy and the safety of R-CHOP in combination with ibrutinib for 6 cycles followed by ibrutinib maintenance for 18 months in ABC-DLBCL patients achieving at least a PR after the induction phase

DETAILED DESCRIPTION:
Step 1 - Screening phase If central review will confirm and define the diagnosis of ABC-DLBCL according the COO, eligible patients will have to sign an additional informed consent prior to receive the study subsequent treatment.

Step 2 - study treatment phases Induction phase: 5 courses of R-CHOP every 21 days combined with ibrutinib (560 mg/day, continuously).

Maintenance phase: patients achieving a CR or a PR after 5 courses of RI-CHOP21 will enter the maintenance phase with ibrutinib (560 mg/day, continuously) for 18 months.

Radiotherapy could be delivered as consolidation treatment at the end of R-chemotherapy, according to Institution local clinical practice, in patients with focal PET positive residual disease and to bone extranodal lesions or scrotum, if testicular involvement irrespective of initial tumor diameter.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically confirmed DLBCL not otherwise specified (NOS). Patients with follicular lymphoma IIIB and large B-cell lymphoma with IRF4 rearrangement can be also included.
* ABC type defined by Lymph2Cx on the NanoString platform. Note: A formalin fixed paraffin embedded lymph node or tumor biopsy specimen must be submitted to Central Pathology for review during the Screening Period. The specimen must have been acquired by a surgical incision or excision biopsy or from a core needle biopsy
* Previously untreated disease
* Age ≥ 18 and < 65 years
* IPI score ≥ 2
* Ann Arbor stage II-IV disease
* Measurable disease ≥ 1.5 cm in longest diameter, and measurable in 2 perpendicular dimensions
* Normal blood count as defined as: absolute neutrophil count ≥1.0 × 10 9 /L independent of growth factor support, platelet count ≥ 100,000/mm 3 or ≥ 50,000/mm 3 if bone marrow (BM) involvement independent of transfusion support in either situation Normal organ functions defined as: creatinine ≤2 times the upper limit of normal (ULN) or estimated Glomerular Filtration Rate (Cockroft-Gault) ≥40 ml/min/1.73m 2 , aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3× the ULN; total bilirubin ≤ 1.5 × the ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN; International normalized ratio (INR) < 1.5 × the ULN in the absence of therapeutic anticoagulation; partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) < 1.5 × the ULN in the absence of a lupus anticoagulant
* Patients with occult or prior hepatitis B infection (defined as HBsAg negative, anti-HBs positive and /or anti-HBc positive) may be included if hepatitis B virus (HBV) DNA is undetectable. These patients must be willing to undergo bi-monthly DNA testing and they should receive prophylaxis with Lamivudine
* No active hepatitis C virus (HCV) infection
* Known availability of biopsy material
* No Central Nervous System (CNS) disease (meningeal and/or brain involvement by lymphoma)
* Absence of active infections
* No peripheral neuropathy or active neurological non-neoplastic disease of CNS
* No major surgical intervention prior 3 months to enrolment if not due to lymphoma and/or no other disease life-threatening that can compromise chemotherapy treatment
* Patient with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study.
* No previous malignancies or patient with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study or patients with any other malignancy in remission without treatment for at least 5 years prior to enrolment
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. - Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [Beta-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Life expectancy > 6 months
* Written informed consent from the patient stating understanding of the purpose and procedures required by the study and willingness to take part in the study

EXCLUSION CRITERIA

* DLBCL including High grade B-cell Lymphomas, both with double hit and NOS according to the 2017 Revised WHO Classification of Tumour of Haematopoietic and Lymphoid Tissues
* GCB-DLBCL after centralized COO profiling
* Any other histologies than DLBCL: composite or transformed disease.
* Primary mediastinal lymphoma (PMBL)
* Known central nervous system lymphoma
* Primary testicular lymphoma
* Any prior lymphoma therapy
* Contraindication to any drug in the chemotherapy regimen
* Left ventricular ejection fraction (LVEF) < 50%
* Neuropathy ≥ grade 2
* Seropositive for or active viral infection with HBV
* HBsAg positive
* HBsAg negative, anti-HBs positive and/or anti-HBc positive with detectable viral DNA
* Known seropositive active HCV
* Human immunodeficiency virus (HIV) infection
* Any of the following abnormal laboratory values (unless any of these abnormalities are due to underlying lymphoma): creatinine ≥ 2 times the ULN (unless creatinine clearance normal, or calculated creatinine clearance < 40 mL/min (using the Cockcroft-Gault formula); AST or ALT ≥3 × the ULN; total bilirubin >1.5 × the ULN: patients with documented Gilbert disease may be enrolled if total bilirubin is ≤ 3.0 × the ULN; INR > 1.5 × the ULN in the absence of therapeutic anticoagulation; PTT or aPTT > 1.5 × the ULN in the absence of a lupus anticoagulant"
* History of stroke or intracranial hemorrhage within the past 6 months.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Any uncontrolled active systemic infection requiring intravenous (IV) antibiotics
* Major surgical intervention prior 4 weeks to enrollment if not due to lymphoma and/or other disease life-threatening that can compromise chemotherapy treatment
* Prior malignancies other than lymphoma in the last 5 years with exception of currently treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix
* Any other medical or psychological condition that might preclude participation in the study or impair the patient's ability to give informed consent.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.
* If female, the patient is pregnant or breast-feeding

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-07-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (1st time point of assessment) | Time between the date of enrolment and the date of disease progression, relapse or death from any cause (24 months)
  PFS of the high/high-intermediate risk patients from date of enrolment
Progression-free survival (PFS) (2nd time point of assessment) | Time between the date of enrolment and the date of disease progression, relapse or death from any cause (36 months)
  PFS of the high/high-intermediate risk patients from date of enrolment
Progression-free survival (PFS) (3dr time point of assessment) | Time between the date of enrolment and the date of disease progression, relapse or death from any cause (48 months)
  PFS of the high/high-intermediate risk patients from date of enrolment

SECONDARY OUTCOMES:
Overall Survival (OS) | Time between the date of enrolment and the date of death from any cause (24, 36 and 48 months).
  Overall Survival
Complete response and Overall Response (CR+PR) rate at the end of induction | End of induction (EOI) (4 months)
  Complete response and Overall Response
Duration of response (DOR) | From the date when criteria for response are met (CR or PR) until the date of progression or relapse. Patients without relapse or progression or death from other causes will be censored at their last assessment date (24 months from response date)
  Duration of response
Complete remission (CRR) after ibrutinib maintenance | End of treatment (EOT) (up to 24 months)
  Complete remission after ibrutinib maintenance
Event Free Survival (EFS) | From the date of enrolment to the date of disease progression, relapse from CR, initiation of subsequent systemic anti-lymphoma therapy after the least 6 cycles of RI-CHOP (each cycle is 21 days), or death whichever occurs first (24, 36 and 48 months)
  Event Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Martelli, Prof., Principal Investigator — Dipartimento di Medicina Traslazionale e di Precisione, Università 'La Sapienza'
Locations (39):
- Italy (39):
  - Ospedale di Castelfranco Veneto - Oncoematologia IOV, Castelfranco Veneto, Treviso
  - A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia, Alessandria
  - Università Politecnica delle Marche- Clinica di Ematologia, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - Centro Riferimento Oncologico- S.O.C. Oncologia Medica A, Aviano
  - IRCCS Istituto Tumori Giovanni Paolo II - U.O.C Ematologia, Bari
  - ASST Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Businco - SC Ematologia e CTMO, Cagliari
  - Arnas Nuovo Ospedale Garibaldi Nesima - U.O.C. Ematologia, Catania
  - Azienda Ospedaliera Universitaria Careggi - Unità funzionale di Ematologia, Florence
  - Ospedale Policlinico San Martino S.S.R.L- IRCCS per l'Oncologia - Ematologia, Genova
  - Azienda Ospedali Riuniti Papardo-Piemonte - S.C. Ematologia, Messina
  - Istituto Scientifico San Raffaele - Unità Linfomi - Dipartimento Oncoematologia, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano - Ematologia, Milan
  - IEO Istitito Europeo di Oncologia - Divisione Ematoncologia, Milan
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Milan
  - Azienda Ospedaliero-Universitaria Policlinico di Modena - Ematologia, Modena
  - Monza - Fondazione IRCCS San Gerardo dei Tintori - Ematologia, Monza
  - Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale - UOC Ematologia Oncologica, Napoli
  - AOU Maggiore della Carità di Novara - SCDU Ematologia, Novara
  - I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1, Padua
  - IRCCS Policlinico S. Matteo di Pavia - Div. di Ematologia, Pavia
  - P.O. Spirito Santo di Pescara - UOS Dipartimentale - Centro di diagnosi e Terapia dei linfomi, Pescara
  - Ospedale Guglielmo da Saliceto - U.O.Ematologia, Piacenza
  - AOU Pisana - U.O. Ematologia, Pisa
  - A.O.R. "San Carlo" - U.O. Ematologia, Potenza
  - Ospedale delle Croci - Ematologia, Ravenna
  - Azienda Unità Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova - Ematologia -, Reggio Emilia
  - Ospedale degli Infermi di Rimini - U.O. di Ematologia, Rimini
  - Dipartimento di Medicina Traslazionale e di Precisione, Università 'La Sapienza', Roma
  - Università Cattolica S. Cuore - Ematologia, Roma
  - Casa Sollievo della Sofferenza - UO Ematologia, San Giovanni Rotondo
  - A.O. S. Maria di Terni - S.C. Oncoematologia, Terni
  - A.O.U. Citta della Salute e della Scienza di Torino - Centro Ematologia Universitaria, Torino
  - A.O.U. Citta della Salute e della Scienza di Torino - S.C.Ematologia, Torino
  - A.O. C. Panico - U.O.C Ematologia e Trapianto, Tricase
  - Azienda Sanitaria Universitaria Integrata Trieste (ASUITS) SC Ematologia, Trieste
  - Ospedale Azienda Sanitaria Universitaria Integrata di Udine (A.S.U.I. Udine)-SOC Clinica Ematologica, Udine
  - Ospedale di Circolo U.O.C Ematologia, Varese

IPD SHARING:
Plan to Share IPD: No